CLINICAL TRIAL: NCT06445894
Title: Accelerated Intermittent Theta-burst Stimulation to Modify Cognitive Function and Balance in Dementia and Memory Loss
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Aimee Nelson, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17300
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Dementia Alzheimers
Keywords: neuroplasticity; transcranial magnetic stimulation; dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active rTMS to M1 (Active Comparator): iTBS will be delivered using a Magstim Rapid 2 stimulator (Magstim, Whitland, UK) guided with neuronavigation (Brainsight, Rogue Research, Montreal, QC, Canada) to target M1. Participants will receive 14 days of stimulation. During each treatment day, three iTBS sessions separated by 15-minute intervals will be delivered. Each iTBS session consists of 600 stimuli delivered in 50 Hz bursts of 3 pulses at 70% of the resting motor threshold. In total, individuals will receive 1800 stimuli delivered each day as performed elsewhere . Following iTBS individuals will participate in 10 minutes of balance training performed on balance board (BTracks https://balancetrackingsystems.com).
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation
- Active rTMS to DLPFC (Active Comparator): iTBS will be delivered using a Magstim Rapid 2 stimulator (Magstim, Whitland, UK) guided with neuronavigation (Brainsight, Rogue Research, Montreal, QC, Canada) to target DLPFC. Participants will receive 14 days of stimulation. During each treatment day, three iTBS sessions separated by 15-minute intervals will be delivered [13,22]. Each iTBS session consists of 600 stimuli delivered in 50 Hz bursts of 3 pulses at 70% of the resting motor threshold. In total, individuals will receive 1800 stimuli delivered each day as performed elsewhere [13,23,27]. Following iTBS individuals will participate in 10 minutes of balance training performed on balance board (BTracks https://balancetrackingsystems.com).
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation
- Placebo rTMS to M1 (Placebo Comparator): sham iTBS will be delivered using a Magstim Rapid 2 stimulator (Magstim, Whitland, UK) guided with neuronavigation (Brainsight, Rogue Research, Montreal, QC, Canada) to target M1. Participants will receive 14 days of placebo stimulation. Following sham iTBS individuals will participate in 10 minutes of balance training performed on balance board (BTracks https://balancetrackingsystems.com).
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Active Repetitive Transcranial Magnetic Stimulation — rTMS is a non-invasive, non-painful procedure used to relieve chronic pain and promote short-term changes. The first dorsal interossesous (FDI) muscle of the left motor cortex will be targeted using neuronavigation software.
  Arms: Active rTMS to DLPFC; Active rTMS to M1
Device: Sham Repetitive Transcranial Magnetic Stimulation (rTMS) — A sham coil will be utilized for the sham rTMS condition. It is important to note that from the participant perspective, the sham stimulation will feel and sound identical to active. The location and all other parameters of Sham rTMS will be identical to Active rTMS.
  Arms: Placebo rTMS to M1

SUMMARY:
The process of aging is accompanied by normal deterioration of body systems, leading to a decline in various functional domains including cognitive, visual, vestibular, somatosensory, and motor function. With this functional decline, there is an increasing burden of care due to the rise of injury, direct and indirect healthcare costs, and the loss of independence in performing daily activities. Notably, falls in the older population represents one of the greatest costs incurred by Canadians annually.

The study investigates whether rTMS delivered to M1 will lead to greater improvement in balance compared to rTMS delivered to DLPFC. Determining this answer will allow greater success in TMS target refinement. Given the profound burden that geriatric medicine has on the Canadian healthcare system, understanding the link between balance and cognition can significantly impact the approach to management of this population.

DETAILED DESCRIPTION:
Approximately 20-30% of Canadian adults >65 years old experience falls each year, and this rate drastically increases for those >85 years of age [2]. With the aging population, the number of annual reported falls has increased by 47% from 2008 to 2020 [3]. Individuals with cognitive impairment exhibit an 8x higher risk of falls compared to those without [4]. Balance is a key risk factor for falls [5-7], and there is evidence suggesting that balance control is a marker of cognitive decline [8]. For example, cognitive function is significantly correlated with postural control [9] and postural sway [10]. In Parkinson's disease, balance has been linked to greater executive dysfunction and slower processing speed [11].

Synaptic plasticity induced via neuromodulatory techniques can lead to improvements in motor and cognitive function. One such technique is Transcranial magnetic stimulation (TMS), a non-invasive form of neuromodulation. To induce synaptic plasticity, magnetic stimuli are delivered via TMS in theta-burst patterns. This includes continuous theta burst stimulation (cTBS) that induces long term depression (LTD)-like changes in neuronal excitability and intermittent theta burst stimulation (iTBS) that induces long term potentiation (LTP)-like changes in neuronal excitability [12]. Previous literature suggests that iTBS may be an effective tool for modulating cognition and motor function.

Wu et al. (2022) found an improvement in memory function of Alzheimer disease patients following a 14-day course of iTBS delivered to the dorsolateral prefrontal cortex (DLPFC) [13]. Trung et al. (2019) showed that 3 days of iTBS delivered to the DLPFC led to cognitive improvements in a sample of Parkinson's disease patients with mild cognitive impairment (MCI) [14]. Regarding balance, iTBS has been shown to be an effective intervention for balance recovery when delivered to the cerebellum [16,17] or the primary motor cortex (M1) [16]. Improvements in gait performance have also been seen following other patterns of stimulation including repetitive TMS (rTMS) in the post-stroke population [18-20]. These improvements in cognition and balance following iTBS may be linked to plastic changes in neuronal structure, as seen in animal models [21].

Accelerated intermittent theta-burst stimulation (iTBS) encompass multiple sessions of iTBS administered within a singular day over the course of several days, consequently diminishing the duration of the treatment regimen. aiTBS has been shown to be a tolerable and safe form of non-invasive brain stimulation with rapid antidepressant efficacy and anti-suicidal effects in patients with major depressive disorder [22-27]. Previous studies have demonstrated aiTBS paradigm which consisted of iTBS delivered 3 times per day separated by 15 min intervals, over the course of 14 days, resulted in an improvement in memory function in individuals with Alzheimer disease [13, 27].

For this study question we have chosen two different stimulation sites. DLFPC is known for its contributions to learning and memory. Individuals with dementia typically receive rTMS stimulation to DLPFC to explore whether cognitive function can be improved (Wu et al., 2020). It has been seen that individuals with dementia suffer from a greater number of falls, it is unclear whether rTMS to DLPFC will improve balance performance and risk of falls better than rTMS delivered to M1, a typical site of stimulation for balance related studies. iTBS has been shown to be an effective intervention for balance recovery when delivered to the primary motor cortex (M1) (Liao et al., 2024). Improvements in gait performance have also been seen following other patterns of stimulation including repetitive TMS (rTMS) in the post-stroke population when delivered to M1 (Wang et al., 2012; Wang et al., 2019; Rastgoo et al., 2016). These improvements in cognition and balance following iTBS may be linked to plastic changes in neuronal structure, as seen in animal models (Tsang et al., 2021).

We there ask the study question whether rTMS delivered to M1 will lead to greater improvement in balance compared to rTMS delivered to DLPFC. Determining this answer will allow greater success in TMS target refinement. Given the profound burden that geriatric medicine has on the Canadian healthcare system, understanding the link between balance and cognition can significantly impact the approach to management of this population

ELIGIBILITY:
Inclusion Criteria:

1. Individuals must be diagnosed with Dementia and/or memory loss by a clinician.
2. Individuals must exhibit adequate oral communication skills and cognitive function sufficient to obtain a score ranging between 10-27 on the Mini-Mental State Exam (Wu et al., 2022).
3. Instructions will be delivered in English; therefore participants must demonstrate an understanding of instruction provided in English or have a caregiver present who can translate and be presented during all study sessions.
4. Individuals must be able to walk or stand with or without personnel or assistive devices.
5. Individuals must be greater than or equal to 50 years of age.

Exclusion Criteria:

* 1. Contraindications to rTMS; presence of a pacemaker, metal/electrical/magnetic implants not including titanium, known history of untreated or uncontrolled psychological disorders, pregnancy, history of seizure or diagnoses of epilepsy, are taking any prescription medications that increase the risk of seizure.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Time Up & Go (TUG) task | At baseline 1-2 days pre-intervention, and 1-2 days post-intervention
  Patients wear their regular footwear and can use a walking aid, if needed. It will begin by having the patient sit back in a standard armchair and identify a line 3 meters, or 10 feet away, on the floor. The participant will be instructed "When I say "Go," I want you to: 1. Stand up from the chair. 2. Walk to the line on the floor at your normal pace. 3. Turn. 4. Walk back to the chair at your normal pace. 5. Sit down again." During this task, IMU will be worn on the ankle to collect movement kinematics relating to balance. During this task two research personnel, one positioned on either side of the participant, will be present in order to stabilize the participant in the case of a loss of balance. In addition, foam padding will be positioned surrounding the patient during standing assessments and moved alongside the patient in walking assessments

SECONDARY OUTCOMES:
Activities-Specified Balance Confidence (ABC) scale | At baseline 1-2 days pre-intervention, and 1-2 days post-intervention
  A patient-reported questionnaire regarding balance confidence during 16 everyday activities. The ABC scale is quick and easy to administer and has demonstrated good reliability, validity, and sensitivity
Mini-Balance Evaluation Systems Test (M-BESTest) | At baseline 1-2 days pre-intervention, and 1-2 days post-intervention
  A sensitive, reliable, valid, and sensitive 14-item scale that assesses dynamic balance [30]. It includes components evaluating anticipatory postural adjustments, responses to perturbation, sensory orientation and dynamic stability during gait. The total score ranges from 0 ("no balance") to 28 ("complete balance"). Each task on the M-BESTest will be scored from 0-2, which correspond to normal, moderate or severe inability to perform the task. In order to complete this test Temper® foam (4 inches thick, medium density T41 firmness rating), chair without arm rests or wheels, incline ramp, stopwatch, a box (9" height) and a 3-meter distance measured out and marked on the floor with tape [from chair] will be required.
Balance Assessment test | At baseline 1-2 days pre-intervention, and 1-2 days post-intervention
  Assesses the capacity of an individual to control center of gravity (COG) within their base of support. While standing on a force platform, subjects are asked to move a cursor indicating their COG from a center target to a peripheral target and back as quickly as possible while minimizing deviation. The process is repeated three times for each of nine peripheral targets in a random order with 30 second rests between each target presentation. Outcome measures derived from the test include movement reaction time (RT) movement velocity (MV), maximum COG excursion (ME), end point COG excursion (EE), and directional control (DC). These LS measures are all impaired in fallers compared to non-fallers [32].
Geriatric Anxiety Inventory (GAI) | At baseline 1-2 days pre-intervention, and 1-2 days post-intervention
  The GAI is a 20-item scale that screens for anxiety symptoms in adults aged 50 and over. It is designed to assess anxiety symptoms over the past week.
Cornell Scale for Depression in Dementia (CSDD) | At baseline 1-2 days pre-intervention, and 1-2 days post-intervention
  The CSDD is a valid screening tool for depression in elderly individuals with and without dementia [34]. This is a 19-item scale that it's designed to assess depressive symptoms over the past week and is completed by the individual's appointed caregiver.
Associative memory | At baseline 1-2 days pre-intervention, and 1-2 days post-intervention
  Associative memory will be assessed using a face-word association task adapted from Wu et al. [13]. In this task, participants will be presented with 12 different pictures of human faces for 12s each. With each face, a common word will be presented, making a face-word pair. The participants will be instructed to memorize the face-word pairs. After a one-minute break, participants were again showed the same faces in a randomized order without the associated word. Participants were asked to recall the unique common word that was presented with each face. The number of successful answers will be summed as the associative memory score. Participants repeated this task twice, with a three-minute interval between each attempt. The average score of the two trials was used as the final associative memory score.
Montreal Cognitive Assessment (MOCA) | At baseline 1-2 days pre-intervention, and 1-2 days post-intervention
  The MOCA is a tool used to assess cognitive impairment [35]. It assesses various aspects of cognition including executive function, memory, language, attention, and orientation. A score less than 25 out of 30 is considered significant for MCI.
Frequency of Falls | At baseline 1-2 days pre-intervention, 6 months post-intervention
  Frequency of Falls: This questionnaire is composed of a single question that asks the number of falls experienced in the past 6 months. In the event that the SDM provides consent, they will be asked for a response to this questionnaire. In the event that the participant provides direct consent they will be asked to answer the question posed on the questionnaire. The researcher will additionally reach out to the family member/caregiver identified on the assent form to acquire this information. In the case of discrepant responses between the participant and the family member/caregiver we will use the response provided by the latter.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster Unviersity, Hamilton, Ontario, Canada